CLINICAL TRIAL: NCT02404896
Title: Expanded-Access for the Use of Metreleptin in Patients With Partial Lipodystrophy Associated With Diabetes Mellitus or Hypertriglyceridemia
Brief Title: Expanded Access Metreleptin Study
Status: Available | Type: Expanded Access
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elif Oral, Professor, Internal Medicine, University of Michigan
Other Study IDs: HUM00094843
Record Dates: First submitted 2015-01-20; First posted 2015-04-01 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Familial Partial Lipodystrophy
MeSH Terms: conditions — Lipodystrophy, Familial Partial | interventions — metreleptin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Metreleptin — Metreleptin open-label treatment
  Other Names: MyaLept

SUMMARY:
Metreleptin was approved in the United States as adjunct to diet as replacement therapy to treat the complications of leptin deficiency in patients with congenital or acquired generalized lipodystrophy in February 2014. The approval was based on results obtained in 2 open-label, investigator-sponsored studies (Studies 991265 and 20010769) conducted at the National Institutes of Health (NIH) to evaluate the safety and efficacy of metreleptin treatment in patients with lipodystrophy and 1 treatment IND (FHA101/MB002-002/MB002-002) conducted by Bristol-Myers Squibb on behalf of AstraZeneca (BMS/AZ) in patients with diabetes mellitus and/or hypertriglyceridemia related to lipodystrophy. These studies enrolled patients with lipodystrophy including both generalized and partial lipodystrophy. Although the marketing authorization restricted the indication to patients with generalized lipodystrophy, meaningful clinical benefit was achieved in a subset of patients with partial lipodystrophy, and these patients from FHA101/MB002-002 form the basis of the request for ongoing treatment under expanded access.

DETAILED DESCRIPTION:
Leptin is a naturally occurring hormone and an important regulator of energy homeostasis and other diverse physiological functions. Circulating levels of leptin closely correlate with the amount of adipose tissue present. Metreleptin, a recombinant analogue of human leptin, is a 147-amino acid polypeptide that differs from the human leptin sequence by 1 additional amino acid, methionine, located at the amino-terminal end. Metreleptin has the same physiological effects as leptin, including regulation of energy homeostasis and metabolic function.

The patient group covered under this expanded access submission has demonstrated evidence of clinical benefit from treatment with metreleptin in clinical study FHA101/MB002-002, and needs expanded access to continue treatment without interruption.

New enrollment, subject to approval by the FDA, can be considered on a case-by-case basis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   a) Before any program procedures are performed, the details of the program will be described to the patient and the patient will be given a written informed consent document to read. If the patient agrees to participate in the program, consent will be indicated by signing and dating of the informed consent document in the presence of program personnel.
2. Target Population

   1. Ability to comply with visits and procedures required by program
   2. Previously enrolled in study FHA101/MB002-002
   3. Has physician-confirmed partial lipodystrophy and had evidence of benefit with metreleptin treatment based on the following metabolic criteria demonstrated within the last year of metreleptin treatment (if on treatment over 1 year) from baseline values:

      * TG reduction ≥ 30% OR
      * HbA1c reduction ≥ 1% OR
      * Decrease in insulin requirements ≥ 40% OR
      * Decrease in episodes of pancreatitis OR
      * Improvement in steatohepatitis OR
      * Withdrawal of metreleptin led to marked worsening of metabolic parameters
3. Age and Reproductive Status

   1. Male or female, over the age of 6 months
   2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the restart of study drug.
   3. Women must not be breastfeeding
   4. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with metreleptin plus 5 half-lives of metreleptin plus 30 days (duration of ovulatory cycle) for a total of 6 months post-treatment completion.
   5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with metreleptin plus 5 half-lives of the metreleptin plus 90 days (duration of sperm turnover) for a total of 3 months post-treatment completion.

Exclusion Criteria:

1. Target Disease Exceptions

   a) Has acquired lipodystrophy and clinically significant hematologic abnormalities (such as neutropenia and/or lymphadenopathy)
2. Medical History and Concurrent Diseases

   1. Has been diagnosed with generalized lipodystrophy
   2. Has been diagnosed with HIV infection
   3. Has a clinically significant medical condition that could potentially affect the risk/benefit ratio for metreleptin treatment and/or the personal well-being of the patient, as judged by the primary treating physician
   4. Has known infectious liver disease
   5. Has known allergies to E. coli-derived proteins or hypersensitivity to any component of metreleptin treatment
3. Other Exclusion Criteria

   1. Prisoners or patients who are involuntarily incarcerated.
   2. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States